CLINICAL TRIAL: NCT02218749
Title: The Effects of Triaging Patients With Musculoskeletal Disorders Directly to Physiotherapists at Primary Health Care Clinics: a Pilot Study and Randomized Controlled Trial.
Brief Title: Triaging Patients With Musculoskeletal Disorders Directly to Physiotherapists at Primary Health Care Clinics.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Organizational barriers
Sponsor: Göteborg University (Other)
Collaborators: Närhälsan Primary care Research and Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 148611; VGFOUGSB-421881 (Other Grant/Funding Number: FoU primärvård Göteborg och Södra Bohuslän)
Record Dates: First submitted 2014-08-15; First posted 2014-08-18 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Initially triaged to physiotherapist (Experimental): Initially triaged to physiotherapist
  Interventions: Other: Initially triaged to physiotherapist
- Initially triaged to physician (Active Comparator): Initially triaged to physician
  Interventions: Other: Initially triaged to physician

INTERVENTIONS:
Other: Initially triaged to physiotherapist
  Arms: Initially triaged to physiotherapist
Other: Initially triaged to physician
  Arms: Initially triaged to physician

SUMMARY:
The purpose of this study is to determine whether initial triaging to physiotherapists of patients with musculoskeletal disorders who seek health care from primary care clinics affects the patients health and/or health care utilization differently than initial consultation with a general practitioner.

ELIGIBILITY:
Inclusion Criteria:

* seeking primary care clinic for musculoskeletal disorder
* age 16-67 years
* speaks enough Swedish or English to understand the patient information and complete the questionnaires
* triage nurse judges it suitable to triage participant to physiotherapist

Exclusion Criteria:

* has received treatment at the clinic by physician or physiotherapist during the preceding month for the same problem
* seeking for chronic musculoskeletal disorder with unchanged symptoms the latest 3 months and for which the patient has already tried physiotherapy
* seeking for help with medical aids other than crutches
* is in need of home care
* has been included in the study earlier

Ages: 16 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Number of physician visits | 1 year
Change in self-evaluated level of pain latest week (0-10 scale) | 3 months

SECONDARY OUTCOMES:
Number of physiotherapist visits | 1 year
Number of days of sick-leave | 1 year
Number of referrals for external examinations and to specialists | 1 year
Changes in health-related quality of life measured with EQ-5D | 2 weeks
Changes in health-related quality of life measured with EQ-5D | 3 months
Changes in health-related quality of life measured with EQ-5D | 6 months
Changes in health-related quality of life measured with EQ-5D | 1 year
Changes in attitudes regarding responsibility for musculoskeletal disorders measured with ARM scale | 2 weeks
Changes in attitudes regarding responsibility for musculoskeletal disorders measured with ARM scale | 3 months
Changes in attitudes regarding responsibility for musculoskeletal disorders measured with ARM scale | 6 months
Changes in attitudes regarding responsibility for musculoskeletal disorders measured with ARM scale | 1 year
Change in experience of functional difficulty measured with DRI scale | 2 weeks
Change in experience of functional difficulty measured with DRI scale | 3 months
Change in experience of functional difficulty measured with DRI scale | 6 months
Change in experience of functional difficulty measured with DRI scale | 1 year
Risk for developing chronic pain measured with the Örebro Musculoskeletal Pain Screening Questionnaire | 2 weeks
Risk for developing chronic pain measured with the Örebro Musculoskeletal Pain Screening Questionnaire | 3 months
Risk for developing chronic pain measured with the Örebro Musculoskeletal Pain Screening Questionnaire | 6 months
Risk for developing chronic pain measured with the Örebro Musculoskeletal Pain Screening Questionnaire | 1 year
Change in self-evaluated level of pain latest week (0-10 scale) | 2 weeks
Change in self-evaluated level of pain latest week (0-10 scale) | 6 months
Change in self-evaluated level of pain latest week (0-10 scale) | 1 year
Prescriptions för analgesics for the actual musculoskeletal disorder | 2 weeks
  Received any prescriptions. Number of prescriptions. Number of occasions prescriptions were received. Type of prescription(s) received.
Prescriptions för analgesics for the actual musculoskeletal disorder | 3 months
  Received any prescriptions. Number of prescriptions. Number of occasions prescriptions were received. Type of prescription(s) received.
Prescriptions för analgesics for the actual musculoskeletal disorder | 6 months
  Received any prescriptions. Number of prescriptions. Number of occasions prescriptions were received. Type of prescription(s) received.
Prescriptions för analgesics for the actual musculoskeletal disorder | 1 year
  Received any prescriptions. Number of prescriptions. Number of occasions prescriptions were received. Type of prescription(s) received.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Bornhöft, MSc, RPT, Principal Investigator — Göteborg University
Locations (3):
- Sweden (3):
  - Närhälsan Eriksberg Health centre, Gothenburg
  - Närhälsan Biskopsgården Health centre, Gothenburg
  - Närhälsan Kyrkbyn Health centre, Gothenburg

REFERENCES:
- [Derived] Bornhoft L, Thorn J, Svensson M, Nordeman L, Eggertsen R, Larsson MEH. More cost-effective management of patients with musculoskeletal disorders in primary care after direct triaging to physiotherapists for initial assessment compared to initial general practitioner assessment. BMC Musculoskelet Disord. 2019 May 1;20(1):186. doi: 10.1186/s12891-019-2553-9. PMID 31043169